CLINICAL TRIAL: NCT02208973
Title: Randomized, Double Blind, Placebo Controlled, Parallel Groups Study to Assess the Safety, Tolerability and Pharmacokinetic Profile of PBF-680 "After Multiple Oral Doses" in Healthy Volunteers.
Brief Title: Study to Assess the Safety, Tolerability and Pharmacokinetic Profile of PBF-680 After Multiple Oral Doses"
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Palo Biofarma, S.L (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IIBSP-PBF-2014-04; 2014-000425-20 (EudraCT Number)
Record Dates: First submitted 2014-08-04; First posted 2014-08-05 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Asthma
Keywords: Adenosine A1 receptor antagonist; adenosine receptor modulator; Asthma; COPD
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- PBF-680 (5 mg) (Experimental): 5 mg of PBF-680
  Interventions: Drug: PBF-680
- PBF-680 (10 mg) (Experimental): 10 mg of PBF-680
  Interventions: Drug: PBF-680
- PBF-680 (20 mg) (Experimental): 20 mg of PBF-680
  Interventions: Drug: PBF-680
- PBF-680 (40 mg) (Experimental): 40 mg of PBF-680
  Interventions: Drug: PBF-680
- PBF-680 (60 mg) (Experimental): 60 mg of PBF-680
  Interventions: Drug: PBF-680
- Placebo (Placebo Comparator): Comparator to the doses of 5, 10, 20, 40 and 60 mg. ( subjects for each dose level 6 are located to active treatment and two to placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PBF-680 — 5, 10, 20, 40 and 60 mg of PBF-680
  Arms: PBF-680 (10 mg); PBF-680 (20 mg); PBF-680 (40 mg); PBF-680 (5 mg); PBF-680 (60 mg)
Drug: Placebo — placebo for the dose of 5, 10, 20 and 40 mg of PBF-680
  Arms: Placebo

SUMMARY:
To assess the safety and tolerability of five doses of PBF-680 (5 mg, 10 mg, 20 mg, 40 mg and 60mg) after repeated (8 days) single daily oral dose administration in young male and female healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects meeting all the following inclusion criteria at screening visit:

  1. Healthy male or females subjects, 18-45 years (inclusive) of age at the time of enrollment.
  2. Females must be of non-childbearing potential (i.e., surgically sterile) or have to use contraceptive measures (non-hormonal) such as condom, diaphragm or cervical/vault cap with spermicide until 28 days post-administration. Males should agree to abstain from sexual intercourse with a female partner or agree to use a condom with spermicide, in addition to having their female partner use some contraceptive measures until 28 days post-administration.
  3. Clinically acceptable blood pressure and pulse rate in supine and standing position. Blood pressure and pulse will be measured after a minimum of 3 minutes of resting.
  4. Body weight within normal range (Quetelet's index between 19 and 26) expressed as weight (kg) / height (m2).
  5. Able to understand the nature of the study and comply with all their requirements.
  6. Free acceptance to participate in the study by obtains signed informed consent form approved by the Ethics Committee of the Hospital (CEIC).

Exclusion Criteria:

* Subjects meeting any of the following criteria at screening visit will be excluded from entry into the study:

  1. History of serious adverse reactions or hypersensitivity to any drug.
  2. Presence or history of allergies requiring acute or chronic treatment (except seasonal allergic rhinitis).
  3. Background or clinical evidence of chronic diseases.
  4. Acute illness two weeks before drug administration.
  5. Having undergone major surgery during the previous 6 months.
  6. Smokers (refrained from any tobacco usage, including smokeless tobacco, nicotine patches, etc., for 6 months prior to the administration of the study medication.
  7. History of alcohol dependence or drug abuse in the last 5 years or daily consumption of alcohol > 40 g for men or 24 gr/day for women or high consumption of stimulating beverages (> 5 coffees, teas or coca cola drinks/ day) for both sexes.
  8. Abnormal physical findings of clinical significance at the screening examination or baseline which would interfere with the objectives of the study.
  9. Need of any prescription medication within 14 days prior to the administration of the drug and non prescription medication or herbal medicines within 7 days prior to the administration of the drug.
  10. Participation in other clinical trials during the previous 90 days in which an investigational drug or a commercially available drug was tested.
  11. Having donated blood during 4 weeks period before inclusion in the study.
  12. Existence of any surgical or medical condition which might interfere with the absortion, distribution, metabolism or excretion of the drug, i.e. impaired renal or hepatic function, diabetes mellitus, cardiovascular abnormalities, chronic symptoms of pronounced constipation or diarrhea or conditions associated with total or partial obstruction of the urinary tract.
  13. 12 lead ECG obtained at screening with PR ≥ 220 msec, QRS ≥120 msec and QTc ≥ 440 msec, bradychardia (<50 bpm) or clinically significant minor ST wave changes or any other abnormal changes on the screening ECG that would interfere with measurement of the QT interval.
  14. Symptoms of a significant somatic or mental illness in the four week period preceding drug administration.
  15. History of hepatitis HBV and / or HCV and / or positive serology results which indicate the presence of hepatitis B surface antigen and / or detectable HCV ribonucleic acid (RNA).
  16. Positive results from the HIV serology.
  17. Females with positive results from the pregnancy test or breast-feeding.
  18. Clinically significant abnormal laboratory values (as determined by the Principal Investigator) at the screening evaluation.
  19. Positive results of the drugs at screening period or the day before starting treatment period. A minimum list of 6 drugs will be screened for inclusion: Amphetamines, Cocaine, Ethanol, Opiates, Cannabinoids and Benzodiazepines (positive results may be repeated at the discretion of the Principal Investigator).
  20. Known hypersensitivity to the study drug or the composition of the galenical form.
  21. History of psychiatric diseases or epileptic seizures.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-05; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events | from day 0 to day 15
  Vital Signs, ECG recordings, laboratory safety test and phisical examination will be performed

SECONDARY OUTCOMES:
Pharmacokinetic Profile Analysis (Plasma concentrations) | from day 1 to day 8
  * Day 1: baseline [pre-dose], [+10 min], [+20 min], [+40min], [+60min], [+ 1.5h], [+2 h], [+ 2.5 h], [+ 3 h], [+ 4h], [+8h], [+ 12h] and [+16h] post-medication;
  * Days 2 to 7: baseline [daily pre-dose] which corresponds at +24h of previous dose;
  * Day 8: baseline [daily pre-dose], [+10 min], [+20 min], [+40min], [+60min], [+1.5h], [+2 h], [+ 2.5 h], [+ 3 h], [+ 4h], [+8h], [+ 12h] and [+16h] and [+ 24h] post-daily medication (D9).

OTHER OUTCOMES:
Adenosine A1 receptor antagonism activity | day 1 and day 8
Leeds Sleep Evaluation Questionnaire | from day 1 to day 8

CONTACTS AND LOCATIONS:
Overall Officials: Joan Martínez Colomer, MD, Principal Investigator — CIM Sant Pau - IIB Sant Pau
Locations (2):
- Spain (2):
  - CIM-Sant Pau - IIB Sant Pau, HSCSP, Barcelona, Barcelona
  - Palobiofarma S.L. (molecule owner), Mataró, Barcelona

REFERENCES:
- See also: Related Info — http://www.iibsantpau.cat/
- See also: Related Info — http://www.palobiofarma.com/